CLINICAL TRIAL: NCT00004860
Title: A Phase II Study of ORZEL (UFT + Leucovorin) in Elderly (at Least 75 Years Old) Patients With Colorectal Cancer
Brief Title: Fluorouracil-Uracil and Leucovorin in Treating Elderly Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067511; E-1299
Record Dates: First submitted 2000-03-07; First posted 2004-04-12 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Cancer
Keywords: stage III colon cancer; stage IV colon cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Leucovorin; Tegafur

INTERVENTIONS:
Drug: leucovorin calcium
Drug: tegafur-uracil

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of fluorouracil-uracil and leucovorin in treating elderly patients who have metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate of elderly patients with metastatic colorectal cancer treated with fluorouracil-uracil and leucovorin calcium (Orzel). II. Evaluate the toxicity profile of this regimen in this patient population. III. Compare response rates obtained in this study with those observed in recent phase III studies in younger patients.

OUTLINE: Patients receive oral fluorouracil-uracil and oral leucovorin calcium (Orzel) every 8 hours for 28 days. Courses repeat every 35 days in the absence of unacceptable toxicity or disease progression. Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 20-55 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic colorectal adenocarcinoma Measurable disease

PATIENT CHARACTERISTICS: Age: 75 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL AST or ALT no greater than 2.5 times upper limit of normal (ULN) Renal: Creatinine no greater than 1.5 times ULN Other: No serious infection No other serious underlying medical condition that would preclude protocol therapy No known hypersensitivity to fluorouracil-uracil or leucovorin calcium

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 6 months since prior adjuvant immunotherapy for colorectal cancer No concurrent immunotherapy Chemotherapy: At least 6 months since prior adjuvant chemotherapy for colorectal cancer No other concurrent chemotherapy Endocrine therapy: No concurrent hormonal therapy Radiotherapy: See Disease Characteristics At least 6 months since prior adjuvant radiotherapy for colorectal cancer Prior radiotherapy for locally symptomatic disease allowed Surgery: Prior surgery allowed Other: No prior therapy for metastatic disease No other concurrent investigational drugs No concurrent halogenated antiviral agents (e.g., lodenosine, fialuridine, FMAU, emtricitabine, and sorivudine)

Ages: 75 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Dates: Start 2000-10-09 (Actual); Primary Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard S. Hochster, MD, Study Chair — NYU Langone Health
Locations (51):
- United States (49):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Gainsville, Gainesville, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - New England Medical Center Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Veterans Affairs Medical Center - Cleveland, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Sooner State, Tulsa, Oklahoma
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Veterans Affairs Medical Center - Pittsburgh, Pittsburgh, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - Veterans Affairs Medical Center - Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
- Puerto Rico (2):
  - MBCCOP - San Juan, San Juan
  - Veterans Affairs Medical Center - San Juan, San Juan

REFERENCES:
- [Result] Hochster HS, Luo W, Popa EC, Lyman BT, Mulcahy M, Beatty PA, Benson AB. Phase II study of uracil-tegafur with leucovorin in elderly (> or = 75 years old) patients with colorectal cancer: ECOG 1299. J Clin Oncol. 2007 Dec 1;25(34):5397-402. doi: 10.1200/JCO.2006.10.4521. PMID 18048821